CLINICAL TRIAL: NCT04258592
Title: 18F-MFBG PET Imaging of the Norepinephrine Transporter in Neural Crest and Neuroendocrine Tumors: a Phase I PET/CT Study
Brief Title: 18F-MFBG PET Imaging of the Norepinephrine Transporter in Neural Crest and Neuroendocrine Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S63142
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Neural Crest Tumor; Neuroendocrine Tumors
Keywords: PET/CT; norepinephrine transporter imaging; 18F-MFBG
MeSH Terms: conditions — Neural crest tumor; Neuroendocrine Tumors | interventions — 3-fluorobenzylguanidine; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): A single dose of 18F-MFBG will be intravenously injected in 10 patients with neural crest tumors or neuroendocrine tumors. Adult patients will first undergo a dynamic PET scan, followed by whole-body PET/CT scans at various time points for a pharmacokinetics study and efficacy assessment. Pediatric patients will undergo, depending on what is feasible for the child, at least 1 and up to 2 static whole-body PET/CTs. In patients 12 years or older, also a dynamic PET scan can be performed.
  Interventions: Drug: (18F)MFBG; Device: PET/CT; Other: Venous blood samples

INTERVENTIONS:
Drug: (18F)MFBG — One intravenous injection of 4 MBq/kg (adults) One intravenous injection of 2 MBq/kg (minor participants)
  Other Names: 18F-MFBG
Device: PET/CT — Adult patients will undergo a dynamic PET scan for the first 30 minutes, followed by 3 static whole-body PET/CTs at 60 ± 10 min, 120 ± 30 min and 180 ± 30 min post injection. Pediatric patients will undergo, depending on what is feasible for the child, at least 1 and up to 2 static whole-body PET/CTs. In patients 12 years or older, also a dynamic PET scan can be performed.
Other: Venous blood samples — Blood samples will be obtained for laboratory safety evaluation for initial screening and safety evaluation after injection. Furthermore, in patients undergoing a dynamic PET scan venous blood samples will be obtained for metabolite analysis and activity measurements at various time points post injection (5 ± 2 min, 10 ± 5 min, 20 ± 10 min, 40 ± 20 min, 60 ± 30 min and 120 ± 60 min in adult participants; 5 ± 2 min, 10 ± 5 min, 30 ± 15 min, 50 ± 25 min, 90 ± 30 min in minor participants).

SUMMARY:
The aim of this study is to evaluate the potential and feasibility of 18F-metafluorobenzylguanidine (18F-MFBG) positron emission tomography (PET) in patients with neural crest and neuroendocrine tumors.

DETAILED DESCRIPTION:
Ten neural crest tumor or neuroendocrine tumor (NET) patients, with a routine clinical 123I-metaiodobenzylguanidine (123I-MIBG imaging) (planar + single photon emission tomography (SPECT)) performed in the previous six months or scheduled within three months, will undergo a dynamic PET scan for the first 30 minutes, followed by 3 static whole-body PET/CTs up to three hours post injection for a pharmacokinetics study and efficacy assessment of 18F-MFBG in humans. Furthermore, a comparison with 123I-MIBG imaging will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged 1 year or older
* Signed Informed Consent by the participant (adult) or his/her parents or legal guardian (minors)
* Subject is diagnosed with a neural crest tumor or neuroendocrine tumor
* Subject is judged to be in good general condition by the investigator on the basis of medical history, physical examination including vital signs and clinical laboratory tests, besides the diagnosis of a neural crest tumor
* Subject should have a routine clinical 123I-MIBG scintigraphy (planar + SPECT/CT) performed within 6 months prior to the inclusion visit or scheduled within 3 months after the inclusion visit
* Adult female subjects should be post-menopausal or surgically sterile or using effective contraceptive with negative pregnancy test. Minor female participants of childbearing potential that are sexually active should be using effective contraceptive with negative pregnancy test

Exclusion Criteria:

* Subject has a previous or ongoing recurrent or chronic disease, other than a neural crest tumor, at high risk to interfere with the evaluation of the trial according to the judgement of the investigator, e.g. known gastro-intestinal, hepatic, renal, cardiovascular, metabolic or hormonal disease, cancer, major neurological or convulsive disorder or any psychiatric disease
* Subject is currently, or within two weeks prior to the inclusion visit, a user (including ''recreational use'') of any illicit drugs, including cannabis, or has a history of drug or alcohol abuse
* Subject is unable to refrain from smoking more than 10 cigarettes per day during the study
* Subject has had exposure to ionizing radiation (> 1 mSv) in other research studies within the last 12 months
* Subject suffers from claustrophobia or cannot tolerate confinement during PET/CT scanning procedures
* Adult subject cannot lie still for 45 minutes inside the scanner. Minor participant cannot lie still for the duration of at least one whole-body PET/CT, varying from 15 to 30 minutes depending on the length of the child, except for children who will be sedated for one scan
* Subject is unwilling to avoid unusual, unaccustomed, or strenuous physical activity (i.e. weight lifting, running, bicycling) from the time of the selection visit until the final safety telephone follow-up interview
* Subject or his/her parents or legal guardian in case of minors, does not understand the study procedure
* Subject is unwilling or unable to perform all of the study procedures, or is considered unsuitable in any way by the principal investigator.
* Subject is potentially pregnant (serum and urinary hCG test will be performed in women where pregnancy is not excluded) or is breast-feeding
* Subject has recently (< 30 days or 5 times the plasma half-life of the investigated drug, whichever is longest) participated or is simultaneously participating in another prospective interventional clinical trial
* Subject has a history of multiple and/or severe allergies to drugs or food
* Subject underwent surgery between the selection and inclusion visit
* Adult subject is mentally or legally incapacitated

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Confirmation of 18F-MFBG as a hNET imaging agent in patients with neural crest and neuroendocrine tumors. | 20 months
  The primary endpoint will be met if in 8 out of 10 patients, at least 80% of the known positive lesions on 123I-MIBG imaging is visualized.

SECONDARY OUTCOMES:
Normal-organ and tumor uptake of 18F-MFBG as a function of time | 20 months
  Patients will undergo dynamic PET scanning followed by three static whole-body PET/CT scans at different time points post injection. Uptake as a function of time (pharmacokinetics) will be studied using the software package PMOD (PMOD technologies LLC, Zürich, Switzerland). Volumes of interest (VOIs) will be delineated in relevant normal organs and tumor lesions on all PET images and standardized uptake values (SUV) in all these VOIs will be measured to compute normal-organ and tumor uptake as a function of time.
Identify the ideal time point for imaging after 18F-MFBG injection. | 20 months
  Tumor-to-background ratios as a function of time will be measured. The time point resulting in optimal tumor-to-background ratios, taking into account a realistic implementation in clinical practice, will be defined as the ideal time point for imaging.
Safety analysis of 18F-MFBG administration: Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | 20 months
  The impact of 18F-MFBG administration on clinical symptoms and signs and biochemistry values will be evaluated. Baseline values will be recorded and subjects will be assessed clinically and with serial biochemical analysis. Adverse events will be scored according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Assessment of lesion targeting by 18F-MFBG as compared to 123I-MIBG | 20 months
  A lesion-by-lesion analysis (visual and semi-quantitative) will be performed to compare the number of detected lesions using both tracers.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Deroose, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pauwels E, Celen S, Baete K, Koole M, Bechter O, Bex M, Renard M, Clement PM, Jentjens S, Serdons K, Van Laere K, Bormans G, Deroose CM. [18F] MFBG PET imaging: biodistribution, pharmacokinetics, and comparison with [123I] MIBG in neural crest tumour patients. Eur J Nucl Med Mol Imaging. 2023 Mar;50(4):1134-1145. doi: 10.1007/s00259-022-06046-7. Epub 2022 Nov 26. PMID 36435928
- [Derived] Pauwels E, Celen S, Vandamme M, Leysen W, Baete K, Bechter O, Bex M, Serdons K, Van Laere K, Bormans G, Deroose CM. Improved resolution and sensitivity of [18F]MFBG PET compared with [123I]MIBG SPECT in a patient with a norepinephrine transporter-expressing tumour. Eur J Nucl Med Mol Imaging. 2021 Jan;48(1):313-315. doi: 10.1007/s00259-020-04830-x. Epub 2020 May 8. No abstract available. PMID 32385645